CLINICAL TRIAL: NCT06746545
Title: A Prospective, Open-label, Single-arm Phase II Clinical Study of Fruquintinib Combined With S-1 for the Treatment of Metastatic Colorectal Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F+S-1-CRC
Record Dates: First submitted 2024-12-11; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: Fruquintinib+S-1

INTERVENTIONS:
Drug: Fruquintinib+S-1 — Fruquintinib: 5 mg, oral, once daily，2w/1w；Q3W S-1：40-60 mg (dosed according to body surface area), oral，2w/1w；Q3W

SUMMARY:
Exploring the efficacy and safety of fruquintinib combined with S-1 for second-line and beyond treatment in patients with advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand this study and voluntarily sign the informed consent form;
2. Age ≥18 years, gender not limited;
3. Confirmed advanced metastatic colorectal adenocarcinoma by histopathological examination;
4. Patients have previously received at least one line of standard therapy containing fluorouracil, oxaliplatin, and irinotecan, and have progressed or are intolerant.

   * Each line of treatment must include one or more chemotherapy drugs for a duration of ≥1 cycle;
   * Adjuvant/neoadjuvant therapy is allowed. If recurrence or metastasis occurs during or within 6 months after completion of adjuvant/neoadjuvant therapy, it is considered a failure of first-line chemotherapy for progressive disease;
   * Prior use of chemotherapy combined with cetuximab or bevacizumab in antitumor treatment regimens is allowed;
5. At least one measurable lesion (RECIST 1.1 criteria);
6. ECOG performance status 0-1;
7. Expected survival time ≥12 weeks;
8. Within 14 days before enrollment, the function of major organs must meet the following requirements (no use of any blood components and cell growth factors within 14 days before enrollment):

   * Absolute neutrophil count ≥1.5×10^9/L;
   * Platelet count ≥80×10^9/L;
   * Hemoglobin ≥8g/dL;
   * Total bilirubin <1.5 times the upper limit of normal (ULN);
   * ALT and AST <2.5 times ULN (<5 times ULN for patients with liver metastasis);
   * Serum creatinine ≤1 times ULN;
   * Endogenous creatinine clearance rate >50ml/min;
9. Women of childbearing age or men with partners who wish to have children must use effective contraceptive measures;
10. Agree to provide blood samples.

Exclusion Criteria:

1. Have previously received treatment with fruquintinib or other anti-VEGFR (vascular endothelial growth factor receptor) inhibitors such as apatinib, regorafenib, and anlotinib;
2. Have previously received treatment with tegafur;
3. Have participated in another drug clinical trial within four weeks before enrollment and received at least one dose of medication, or have received other systemic antitumor treatments, including chemotherapy, signal transduction inhibitors, hormone therapy, and immunotherapy within four weeks before enrollment;
4. Patients currently have diseases or conditions that affect drug absorption, or patients are unable to orally take fruquintinib;
5. Patients currently have active gastric and duodenal ulcers, ulcerative colitis, and other gastrointestinal diseases, or have active bleeding from unresected tumors, or other conditions that may cause gastrointestinal bleeding or perforation as judged by the investigator;
6. Have active bleeding or bleeding tendencies;
7. Have uncontrollable malignant pleural effusion, ascites, or pericardial effusion (defined as not effectively controlled by diuretics or puncture as judged by the investigator);
8. Have a history of severe cardiovascular and cerebrovascular diseases:

   * Cerebral vascular accidents (except for lacunar infarction, minor cerebral ischemia, or transient cerebral ischemic attacks), myocardial infarction, unstable angina, poorly controlled arrhythmias (including QTc interval for males ≥ 450ms, females ≥ 470ms) (QTc interval calculated using the Fridericia formula) within 6 months before the first dose of the study drug;
   * New York Heart Association (NYHA) heart function classification > II or left ventricular ejection fraction (LVEF) < 50%;
9. Have had other malignancies in the past 5 years, except for skin basal cell or squamous cell carcinoma after radical surgery, or cervical carcinoma in situ;
10. Have clinically uncontrolled active infections, such as acute pneumonia, active hepatitis B or C (history of hepatitis B virus infection not under drug control, HBV DNA ≥1×10^4 copies/mL or >2000 IU/mL);
11. Have clinically symptomatic central nervous system metastases and/or meningeal carcinomatosis;
12. Patients currently have uncontrolled hypertension with medication, defined as: systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg after taking antihypertensive drugs;
13. Urinalysis indicates urinary protein ≥2+, and re-examined 24-hour urinary protein quantity >1.0g;
14. Pregnant (positive pregnancy test before medication) or breastfeeding women;
15. The investigator judges that there are clinically significant severe electrolyte abnormalities, or the investigator believes that the patient is unsuitable for participation in this clinical study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks, until the occurrence of progressive disease (PD), using RECIST v 1.1

SECONDARY OUTCOMES:
Objective response rate (ORR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Overall survival (OS) | from randomization until death due to any cause, assessed up to 3 year
  Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD).
Disease control rate (DCR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year]
  Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD),using RECIST v 1.1
Safety and tolerance evaluated by incidence, severity and outcomes of AEs | from first dose to 30 days post the last dose
  Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 5.0

OTHER OUTCOMES:
Exploratory study endpoints. | Perform ctDNA tests on patients' blood at the start, after the first three cycles of treatment, and when disease progresses,from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Circulating Tumor DNA (ctDNA) changes.

IPD SHARING:
Plan to Share IPD: Undecided